CLINICAL TRIAL: NCT07168707
Title: A Culturally Adapted Group-Based, Emotional Awareness and Expression Therapy Intervention - Hebrew (EAET-H) for Chronic Pain Patients Treated With Medical Cannabis in Israel - A Pilot Study
Brief Title: Culturally Adapted EAET-H for Chronic Pain Patients Using Medical Cannabis in Israel - A Pilot Study
Acronym: EAET-H
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Reuth Rehabilitation Hospital (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0017-21-RRH
Record Dates: First submitted 2025-08-16; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Chronic Musculoskeletal Pain; Cannabis Use
Keywords: Chronic musculoskeletal pain; Cannabis Use; Emotional Awareness and Expression Therapy; Emotional Therapy; Psychological Therapy; Group-Based

STUDY DESIGN:
Intervention Model Description: A single-arm pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group-based Emotional Awareness & Expression Therapy - Hebrew (EAET-H) (Experimental): This pilot study will use the eight-session group EAET manual developed by Mark A. Lumley and Howard Schubiner. Several adaptations to this manual were made: a) Manual's translation to the Hebrew language; b) Adaptations to the Israeli context and setting; c) Manual's language was changed from "fibromyalgia" to "chronic pain" and adaptations were made accordingly. Group participants will receive a class syllabus and an educational booklet of the EAET approach. Each group meeting will be led by two instructors, a psychologist and a physiotherapist.
  Interventions: Other: Group-based Emotional Awareness & Expression Therapy - Hebrew

INTERVENTIONS:
Other: Group-based Emotional Awareness & Expression Therapy - Hebrew — This pilot study will use the eight-session group EAET manual developed by Mark A. Lumley and Howard Schubiner. Several adaptations to this manual were made: a) Manual's translation to the Hebrew language; b) Adaptations to the Israeli context and setting; c) Manual's language was changed from "fibromyalgia" to "chronic pain" and adaptations were made accordingly. Group participants will receive a class syllabus and an educational booklet of the EAET approach. Each group meeting will be led by two instructors, a psychologist and a physiotherapist.
  Other Names: EAET-H

SUMMARY:
The goal of this clinical trial is to evaluate whether a culturally adapted group-based emotional therapy named "Emotional Awareness and Expression Therapy" can help reduce chronic pain and improve emotional well-being in Israeli adults who suffer from chronic musculoskeletal pain and are treated with medical cannabis.

Researchers will compare patients who receive the emotional therapy along with their usual care to patients who receive usual care only, to see if the therapy leads to better outcomes in pain, mental health, and daily functioning.

Participants will attend a weekly 1.5-hour group therapy session for 8 weeks; Take part in group discussions and emotional processing exercises; Complete questionnaires about pain levels, mood, sleep, and quality of life; Continue their usual medical treatment as prescribed by their doctors.

DETAILED DESCRIPTION:
The rising prevalence of chronic pain conditions poses a significant challenge to societies and healthcare systems globally. Despite medical advancements, many individuals continue to face chronic pain daily, with only limited success in alleviating pain and enhancing physical and emotional well-being. Furthermore, the psychological burden associated with chronic pain highlights the critical need for integrating psychological support within chronic pain treatment strategies. Emotional Awareness and Expression Therapy (EAET) has demonstrated considerable reductions in pain and improvements in psychological conditions such as depression and anxiety among adults with various chronic pain types. However, the EAET intervention has never been tested on patients treated with medical Cannabis and has not yet been evaluated in Israel. Furthermore, we propose that adapting the EAET program to reflect local cultural perspectives on pain and its management will be essential for its effective implementation among Israeli patients.

This study aims to culturally adapt the Emotional Awareness and Expression Therapy - Hebrew (EAET-H) eight-session group-based protocol, for Israeli patients with chronic pain receiving medical Cannabis. The study includes a culturally adaptation of the EAET-H according to the steps outlined by Escoffery and colleagues and fidelity assessment through a single-arm pilot trial, which will assess its implementation fidelity, feasibility, acceptability, and preliminary efficacy on pain severity compared to the usual care. The secondary outcome measures that will be assessed in this study are: pain interference and disability, pain catastrophizing, fear and pain believes, mood and satisfaction with life, physical functioning and quality of life, sleep and fatigue, global impression of change, health service utilization and cannabis consumption.

Description of the intervention: An innovative psychological treatment, EAET is a psychotherapeutic approach that emphasizes the role of emotional processing of unresolved trauma, stress and conflict in the treatment of CP and somatic symptoms. The intervention will be delivered as a 1.5-hour weekly group session for a period of 8 weeks. Each session will include two parts, theoretical and practical, and will combine group discussion and sharing experiences.

The study will take place at "Reuth" Rehabilitation Hospital, Tel- Aviv. Chronic musculoskeletal pain patients who are also medical cannabis consumers, treated at the pain and cannabis clinics will be recruited for the study.

Following completion of this research, a well-defined protocol for a group-based EAET program in Hebrew will be developed, tailored to the Israeli context with culture-specific norms and beliefs to effectively meet patients' unique needs. This research aims to provide clear insights into the feasibility and preliminary efficacy of the adapted program through a rigorous pilot trial. This step is marking the first instance this innovative approach, found to be superior to traditional cognitive-behavioural therapy treatments, is tested among pain patients who are treated with medical Cannabis and in Israel. It is expected to significantly reduce pain levels and disability while alleviating the mental strain experienced by patients-areas currently inadequately addressed. The anticipated result is a major advancement in the existing chronic pain treatment paradigm in Israel, incorporating a significant psychological component and capitalizing on the benefits of group therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with any chronic musculoskeletal pain (≥ three months in duration). widespread pain or fibromyalgia or any combination of these conditions;
2. Treated with medical Cannabis;
3. Physical and mental ability to participate in group discussions;
4. Explicitly endorsed an interest in exploring potential emotional factors contributing to their somatic symptoms;
5. Signed informed consent form

Exclusion Criteria:

1. The following conditions will be excluded: confirmed hip/knee osteoarthritis, radiculopathy, electromyography-confirmed "tunnel" syndromes, autoimmune disease that typically generates pain (e.g., rheumatoid arthritis or multiple sclerosis, inflammatory bowel disease, systemic lupus, sickle cell disease), cancer, and chronic infection associated with pain;
2. Severe mental illness or psychiatric disorder such as schizophrenia, bipolar I disorder, multiple personality disorder, or dissociative identity disorder not controlled with medications. In addition, active suicide or violence risk in the past year, active severe alcohol or substance use disorder.
3. Unable to fluently read or converse in Hebrew;
4. Participation in any other clinical study or program focusing on psychological or behavioral intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory (BPI) - 4 items of pain severity | Baseline and after eight weeks
  The BPI is a self-report questionnaire used to evaluate pain severity and includes four items. These items assess the intensity of pain at its worst, least, average, and current levels.

SECONDARY OUTCOMES:
Brief Pain Inventory (BPI) - 7 items of pain interference | Baseline and after eight weeks
  The BPI is a self-report questionnaire used to assess the impact of pain on daily functioning. Its seven pain interference items measure how pain affects activities such as general activity, mood, walking ability, normal work, relations with others, sleep, and enjoyment of life.
The Hospital Anxiety and Depression Scale (HADS) | Baseline and after eight weeks
  The HADS is a 14-item self-report questionnaire designed to assess symptoms of anxiety and depression in non-psychiatric hospital patients. It consists of two subscales-seven items each for anxiety (HADS-A) and depression (HADS-D).
Pain Self-Efficacy Questionnaire (PSEQ) | Baseline and after eight weeks
  The PSEQ is a 10-item self-report tool designed to assess the confidence of individuals with chronic pain in performing daily activities despite their pain.
Pain Catastrophizing Scale (PCS) | Baseline and after eight weeks
  The PCS is a 13-item questionnaire that measures negative thought patterns related to pain. It assesses three components: rumination, magnification, and helplessness. Higher scores indicate greater levels of pain catastrophizing.
Fear-Avoidance Beliefs Questionnaire (FABQ) | Baseline and after eight weeks
  The Fear-Avoidance Beliefs Questionnaire (FABQ) is a self-report tool that assesses the extent to which fear and avoidance beliefs about physical activity and work contribute to a person's chronic pain. It consists of 11 items divided into two subscales: physical activity and work.
The Satisfaction with Life Scale (SWLS) | Baseline and after eight weeks
  The SWLS is a 5-item self-report questionnaire that measures overall life satisfaction.
Toronto Alexithymia Scale (TAS) | Baseline and after eight weeks
  The TAS is a 20-item self-report questionnaire that can be used to identify issues relating to alexithymia, such as difficulty identifying and describing feelings and externally oriented thinking
The Pittsburgh Sleep Quality Index (PSQI) | Baseline and after eight weeks
  The PSQI is a 19-item self-report questionnaire that assesses sleep quality and disturbances over a 1-month period. It yields a global score based on seven components, including sleep duration, latency, and disturbances.
The Fatigue Severity Scale (FSS) | Baseline and after eight weeks
  The FSS is a 9-item self-report questionnaire that measures the impact of fatigue on daily functioning.
The Patient Global Impression of Change (PGIC) | After eight weeks
  The PGIC is a single-item self-report measure that assesses a patient's overall perception of improvement or decline following treatment.
Medical cannabis consumption | Baseline and after eight weeks
  Three questions regarding the frequency of cannabis use and the method of cannabis consumption.
Health care use | Baseline and after eight weeks
  Four questions regarding the medications the patient takes regularly, the treatments they receive and their frequency, and doctor visits within the past three months.

OTHER OUTCOMES:
Acceptability questionnaire | After four weeks and eight weeks
  An acceptability questionnaire was developed specifically for the current study, consisting of eight items assessing the participant's acceptance of the program (e.g., satisfaction, perceived usefulness of the content, etc.).
Feasibility measures - Rates of recruitment | After eight weeks
  Documentation will be kept of participants who were eligible for the study, gave informed consent, and actively participated in the program. The study will be considered feasible if ≥50% of eligible patients will be enrolled in the study.
Feasibility measures - Session attendance | After eight weeks
  A participant's attendance record will be maintained for each session. The study will be considered feasible if the mean attendance at meetings will be ≥6 of the 8 sessions.
Feasibility measures - Retention | After eight weeks
  A record will be created of participants who completed the program and filled out the post-intervention questionnaires. The study will be considered feasible if ≥70% of enrolled participants will complete the post-intervention survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Reuth Rehabilitation Hospital, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
IPD will be shared only with researchers on the study team and not with any individuals outside the team. Additionally, the data will be stored on the computers of the research institute at the hospital where the intervention program is being conducted.

REFERENCES:
- [Background] Lumley M, Ph. Emotional Awareness and Expression Therapy (EAET): A Group-Based Treatment Manual for Patients with Fibromyalgia and Related Centralized Chronic Pain Disorders.
- [Background] Lumley MA, Schubiner H. Psychological Therapy for Centralized Pain: An Integrative Assessment and Treatment Model. Psychosom Med. 2019 Feb/Mar;81(2):114-124. doi: 10.1097/PSY.0000000000000654. PMID 30461545